CLINICAL TRIAL: NCT03172026
Title: Maraviroc to Augment Rehabilitation Outcomes After Stroke
Acronym: MAROS
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Poor recruitment for each site, partly related to Covid epidemic.
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Bruce H. Dobkin, Principal Investigator, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB#16-001733
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Results first posted 2021-08-03 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Stroke
Keywords: Telerehabilitation; Maraviroc
MeSH Terms: conditions — Stroke | interventions — Maraviroc; Rehabilitation

STUDY DESIGN:
Intervention Model Description: We plan a parallel group, randomized controlled pilot trial at 3 sites, UCLA, Yale and Burke Neurological Institute in White Plains, NY, to gather enough entries in a shorter time and to better generalize the results of this phase II/III pilot trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Maraviroc + Augmented Rehabilitation (Experimental): Participants will take Maraviroc 300 mg daily for 60 days, plus receive rehabilitation therapy as prescribed by the doctors and via telerehabilitation.
  Interventions: Drug: Maraviroc 300 mg; Behavioral: Rehabilitation therapy
- Placebo + Augmented Rehabilitation (Placebo Comparator): Participants will take placebo 300 mg daily for 60 days, plus receive rehabilitation therapy as prescribed by the doctors and via telerehabilitation.
  Interventions: Behavioral: Rehabilitation therapy; Drug: Placebo 300 mg

INTERVENTIONS:
Drug: Maraviroc 300 mg — FDA approved chemokine receptor (CCR5) inhibitor. Maraviroc will be started within two weeks of discharge from inpatient rehabilitation, which most often will occur from 4-6 weeks after stroke onset.
  Other Names: Selzentry
  Arms: Maraviroc + Augmented Rehabilitation
Behavioral: Rehabilitation therapy — All participants will have routine outpatient or home health physical and occupational therapy after inpatient discharge as prescribed by their physicians.
  Each group will be contacted weekly by phone to help maintain interest in the trial, count the number of usual care physical and occupational therapy completed, assure use of the assigned medication, ask about possible adverse reactions, and to encourage them to be active. The coordinator will obtain this information and provide the feedback using a standard script and checklist. A unique aspect of this trial is a telerehabilitation component that aims to give feedback to all participants to practice with the affected arm and walk daily.
Drug: Placebo 300 mg — Matched placebo will be started within two weeks of discharge from inpatient rehabilitation, which most often will occur from 4-6 weeks after stroke onset.
  Arms: Placebo + Augmented Rehabilitation

SUMMARY:
After stroke, the combination of progressive skills practice in an adequate dose, exercise for fitness, and reduced sedentary time will augment motor and cognitive outcomes. Sensorimotor and cognitive improvements after stroke often reach a general plateau by approximately 12 weeks after onset, however. Drugs that might enhance learning or neural repair, as well as other molecular and synaptic adaptations that occur during skills training and fitness exercise, might extend that recovery curve, although to date only fluoxetine has given any hint of this. Most trials have tested agents that modulate neurotransmitters. Several very recent preclinical experiments and observational studies in patients after stroke suggest that the commercially available medication, Maraviroc, a CCR5 antagonist, may augment skills learning during rehabilitation training, especially during the first three months after onset, by affecting CREB and synaptic plasticity.

The investigators will carry out a randomized controlled trial of Maraviroc in patients with disabilities severe enough to have required inpatient stroke rehabilitation and, based on our preclinical data, who can start the drug intervention within 6 weeks of stroke onset. The investigators will compare usual post-stroke care plus placebo versus Maraviroc given for 8 weeks in 60 participants. However, to try to maximize the amount of practice that is most relevant to the primary outcome measurements and determine whether or not Maraviroc can enhance the effects of training, as hypothesized, all participants will be tele-monitored by mobile health devices and will receive weekly telephonic encouragement, based on device data, to walk, reduce sedentary time, and reach and grasp in the home in between usual care therapies. Compliance, serial motor changes over time, and self-management skills in making use of the telerehabilitation devices will be a nested substudy of feasibility of remote monitoring and feedback.

DETAILED DESCRIPTION:
Background

After stroke, the combination of progressive skills practice in an adequate dose, exercise for fitness, and reduced sedentary time will augment motor and cognitive outcomes. Sensorimotor and cognitive improvements after stroke often reach a general plateau by approximately 12 weeks after onset, however. Drugs that might enhance learning or neural repair, as well as other molecular and synaptic adaptations that occur during skills training and fitness exercise, might extend that recovery curve, although to date only fluoxetine has given any hint of this. Most trials have tested agents that modulate neurotransmitters. Several very recent preclinical experiments and observational studies in patients after stroke suggest that the commercially available medication, Maraviroc, may augment skills learning during rehabilitation training especially during the first three months after onset, by acting on unique molecular components for novel learning.

The C-C chemokine receptor 5 (CCR5) is a seven-transmembrane G protein-coupled receptor that mediates HIV virus cellular entry. Individuals who are homozygous for a 32 base pair deletion in the CCR5 gene (CCR5D32), and subsequently do not express functional CCR5, are highly protected from infection with R5 HIV-1. The receptor is expressed in microglia, astrocytes and neurons in many regions of the brain. Dr. Alcino Silva at UCLA postulates that this receptor is involved in learning and memory. In a series of elegant experiments, he showed 1) CCR5 deficiency results in enhancements in hippocampal learning and memory and in experience-dependent sensory plasticity; and 2) CCR5 overexpression leads to learning and memory deficits. Decreasing the function of CCR5 increases MAPK/CREB signaling, long-term potentiation, hippocampus-dependent memory, and neocortical experience-dependent plasticity. Ligand binding to CCR5 is known to modulate several parallel signaling cascades implicated in learning and memory, including the suppression of adenyl cyclase, as well as the activation of the PI3K/AKT and P44/42 MAPK signaling. These findings support the application of brain permeable CCR5 antagonists, not only as a combination drug in antiretroviral therapy, but also as a treatment for cognitive deficits caused by HIV. In addition, the studies suggest that the receptor is a novel target to augment learning and memory in those with cognitive and motor deficits in relation to training.

Several preclinical models of stroke and traumatic brain injury from Drs. ST Carmichael, Alcino Silva, and Esty Shohami suggest that the FDA-approved CCR5 reversible co-receptor antagonist, Maraviroc, may lead to better motor outcomes when combined with training, presumably due to enhanced learning. Stroke induces CCR5 expression in neurons in the first month after onset in a mouse model (Carmichael). Knockdown of CCR5 in the motor cortex of adult mice improves recovery after stroke (Carmichael and Silva et al). Maraviroc also improves motor recovery in this model. An Israeli post stroke observational trial (TABASCO, Einor Ben Assayag, et al.) enabled a test of the effects of a naturally occurring loss of function mutation in CCR5 (CCR5 delta32). About 15% of the Ashkenazi Jewish population carries the deletion (CCR5 rs333 - 32). This group in TABASCO had better outcomes for walking speed and the Berg Balance Scale. A Washington University observational study that included some subjects with this deletion also looked positive for better outcomes, but was more equivocal, based on differences in stroke type. Neither gene association study has been published yet.

Maraviroc is the only CCR5 antagonist currently approved by the United States Food and Drug Administration, the European Commission, Health Canada. Maraviroc (Selzentry, Pfizer) is a small molecule currently approved for treatment of patients infected with R5-tropic HIV-1. It is metabolized by CYP3A4. The dose may have to be adjusted when given with CYP3A4 inducers or inhibitors, primarily drugs that are also used for HIV therapy, but also for several anticonvulsants. None of the subjects in the proposed trial will be entered if on these medications. The drug has a good pharmacokinetic profile with relatively low protein binding and high bioavailability when given at standard doses twice a day. It is moderately lipophilic, so it can penetrate the blood-brain barrier. At a single dose of 300 mg, time to maximum concentration occurred by two hours post-treatment in humans. The terminal half-life is 14-18 hours, so a single dose used during the time of training in the proposed protocol should be adequate, rather than the BID treatment for AIDS. Despite low CSF concentrations, the drug suppresses CSF viral load. It potently inhibits downstream CCR5 signaling and does not induce CCR5 internalization, suggesting that the drug is a functional CCR5 antagonist.

Aims

Given the potential for Maraviroc to augment rehabilitation training, the investigators will carry out a trial of Maraviroc in patients with disabilities severe enough to have required inpatient stroke rehabilitation and, based on our preclinical data, who can start the drug intervention within 6 weeks of stroke onset. The stud design is a parallel group, randomized controlled pilot trial at 3 sites, the Department of Neurology at the UCLA (Bruce Dobkin, MD), the Burke Neurological Institute in White Plains, NY, (Tomoko Kitago, MD) and the Department of Neurology at the Yale University (Lauren Sansing, MD) to gather enough entries in a shorter time and to better generalize the results of this phase II/III pilot trial. Usual post-stroke care plus placebo will be compared to Maraviroc given for 8 weeks in 60 participants (up to 66 to account for dropouts). The primary outcome measurements will be gains in walking and functional use of the affected upper extremity, continuously monitored remotely, as well as formally assessed at 4 and 8 weeks after initiating the drug and at 6 months (primary endpoint) post stroke onset. To try to maximize the amount of practice that is most relevant to the primary outcome measurements and determine whether or not Maraviroc can enhance the effects of training, as hypothesized, all participants will be monitored by mobile health devices and will receive weekly encouragement, based on device data, to walk, reduce sedentary time, and reach and grasp in the home in between usual care therapies. The amount of use of these telerehabilitation devices will be a nested substudy of feasibility.

Hypothesis 1: Subjects who take Maraviroc plus outpatient and home-based rehabilitation therapy managed remotely will improve significantly more in the primary outcomes of walking speed and upper extremity function by the Action Research Arm Test (ARAT) compared to the placebo drug group at the 6-month post stroke assessment.

Hypothesis 2: The feasibility of home-based telerehabilitation practice will be revealed by the finding that at least 75% of all participants will have achieved compliance for at least 150 minutes of walking and 100 minutes of reach and grasp practice weekly.

Methods

Consent Process:

Participants will be identified from the inpatient stroke rehabilitation admissions to the UCLA affiliated California Rehabilitation Institute (CRI) and from referrals to Burke and to Yale. The Burke site will have its own IRB review managed by its PI.

On admission to CRI, patients have the option to sign a consent to be contacted about research projects that might be applicable to them. Potential participants who have signed this will be contacted by a study investigator. In addition, a flyer (submitted) will be provided to patients with stroke during their inpatient rehabilitation stay who may be interested in the study.

Randomization:

Participants will be assigned to the control or experimental group using a 1:1 computer-generated randomized allocation schedule in the REDCap clinical database. Assignment (for both research sites) occurs automatically upon the entry of eligibility criteria.

All members of the research team and the subjects will be blinded as to allocation. The study statistician and the rest of the Safety Committee will have access to the assignment if necessary (e.g., adverse drug reaction).

Each site will enter 20-25 subjects, approximately half into each of the trial arms. Entries will be accomplished within 30 months with follow-up assessments and data analyses by the end of 36 months.

Baseline Studies:

Age, gender, body mass index, ethnicity, living place, work status, caregiver support, date of stroke, date of transfer for inpatient rehabilitation, lesion type (TOAST) and location, personal risk factors for stroke, medications, and FIM for level of pre-stroke walking and ADLs will be collected. Other measures will include the National Institutes of Health Stroke Scale (NIHSS), British Medical Council manual muscle exam for eligibility, motor FIM score, 10-m walking speed, 6-min walking distance, and Action Research Arm Test (ARAT). The investigators will record the average two blood pressures and heart rates on the day of entry and the most recent HbgA1c and lipid panel, liver function tests, creatinine/BUN, and MRI/CT imaging results from the inpatient rehabilitation medical record. If liver function tests or creatinine cannot be found, the tests will be obtained at the outpatient research site as a cost to the study. Drs. Dobkin and Dorsch will review each imaging study to localize the relevant stroke lesion by consensus. An email address and phone number for the patient and a close contact will be kept separate from the clinical database by the coordinator.

Interventions:

Maraviroc: Medications are often in flux during inpatient rehabilitation, so Maraviroc or placebo will be started within two weeks of discharge, which most often will occur from 4-6 weeks after stroke onset. A 1-month supply of capsules will be handed to participants after the Consent has been signed, baseline measurements obtained, and randomization assigned, usually on the same day. The second 1-mo supply will be provided during a scheduled interim measurement assessment at UCLA near the end of the 4th week on medication. Pill counts will be taken on the returned bottle. Participants will take either Maraviroc or a placebo at a dose of 300 mg at 6-8AM. The capsules will be supplied by each site's pharmacy and assigned based on a randomization schema.

Based upon Pfizer's reports on premarketing and post marketing studies of Maraviroc and our review of the literature, no dose adjustment is necessary in patients with even mild-to-moderate renal impairment. The drug does not affect the QT interval. At high doses (600mg or more), it may induce orthostatic hypotension, so it is recommended that users who also take an anti-hypertensive medication be asked about symptoms of orthostatic hypotension. Of note, 8% of patients in active and placebo drug groups described orthostatic symptoms in a large trial. In HIV trials, 1.3% of subjects had cardiovascular events, more than in the placebo group, but the link to the drug was unclear and symptoms occurred only in those with known cardiac disease. Also, no greater incidence of infection, rash or other CNS symptoms was noted in these subjects. An occasional Stevens-Johnson syndrome and drug rash with eosinophilia and systemic symptoms did occur (seen only in post marketing surveillance, not in controlled trials), so complaints of rash, fever, joint or muscle aches, blisters, facial edema, etc. will be part of our weekly phone call surveillance plan. Participants will be told to stop their medication immediately should such symptoms occur and their physician notified. Of note, St John's wort should not be used with the medication since it decreases the concentration of Maraviroc.

The drug is metabolized by the liver, so using it in persons with more than mild hepatic disease, especially in the presence of a CYP3A inhibitor, would have to be closely monitored; our participants will be free of hepatic, as well as renal impairment. The recommendation from the FDA is to obtain liver function tests prior to starting the drug and again should symptoms such as rash or hepatitis occur. This rather rare adverse reaction tends to occur at about one month after starting the medication (in less than 4% on the drug or placebo) , so the investigators will obtain a bilirubin and transaminases at the planned 1-month follow up.

Adverse events related to the medication assignment, to rehabilitation practice or to other causes will be adjudicated by the Safety Committee with input from the PI.

Rehabilitation therapy: All participants will have routine outpatient or home health physical and occupational therapy after inpatient discharge as prescribed by their physicians.

Each group will be contacted weekly by phone to help maintain interest in the trial, count the number of usual care physical and occupational therapy completed, assure use of the assigned medication, ask about possible adverse reactions, and to encourage them to be active. The coordinator will obtain this information and provide the feedback using a standard script and checklist.

A unique aspect of this trial is a telerehabilitation component that aims to give feedback to all participants to practice with the affected arm and walk daily. All participants will be asked to wear a FitBit ankle sensor connected to the cloud. Data includes daily sedentary and active time. At the weekly call, participants will be reminded to try to build up to walking at least 3 times a day for at least 10 minutes per bout and reduce sedentary time. Behavioral modification techniques that the investigators have been using successfully, based on sensor data, will be employed.

Participants will also be given a LEAP Motion Controller device that sits in the bottom of a 12x18" box covered by a clear plastic lid. This simple system enables us to monitor practice of reaching and grasping with the affected upper extremity in the home. At the weekly call, they will be encouraged to perform 20-30 minutes daily of reach, grasp and pinch actions with small common items and practice bringing the affected hand to the mouth. Items will be moved from one corner of the rectangular top to another in a fixed sequence. A unique feature of this trial is that telerehabilitation data will provide ground truth about how much participants practiced, which may enable a dose-response and responder-nonresponder analysis. For example, if a subject is taking the active medication, but never practices, outcomes may be less positive than for the person who does practice as prescribed.

A data manager at UCLA will review all incoming data for completeness and quality as well as ensure proper use of the systems (e.g. make sure devices are charged regularly, automatic data uploads occur without problems, and practice data are processed correctly). All feedback will be provided by the UCLA staff.

Statistical Analyses:

An observational trial (Lohse and Lang, 2016) found that walking speed increases at 0.1m/s per month and the ARAT increases by 2.9 points monthly within the time frame of this trial.

For the walking speed outcome, the evaluable sample size of 30 in each group will have 80% power to detect a difference in means of -0.206 (m/s), the difference between an assumed usual care walking speed of 0.51 (SD=0.28) and an assumed intervention group mean walking speed of 0.716. This assumes a common standard deviation in the two groups and a two group t-test with a 0.05 two-sided significance level. The estimates for the mean and standard deviation for walking speed come from the LEAPS RCT (Duncan, N Engl J Med, 2011). The investigators plan to enroll 66 patients to account for an expected 10% drop-out rate. The t-test used for the power calculation is a simplification of the mixed effects analysis plan for the primary endpoints.

For the ARAT sum score, analysis is based on a statistical power of 80% with an alpha of 5% for detecting a meaningful difference of 6 points, i.e., a 10% change, which has been suggested by several completed trials. In a stroke trial, the standard deviation was 8 points measured at 2 weeks post stroke. Again, a sample size of 60 plus 10% dropout rate should suffice.

Primary Analyses: As appropriate, t-tests, Wilcoxon rank sum, or chi-square tests will be employed to evaluate differences in baseline clinical characteristics between trial participants. Using the mixed effects model for Hypothesis 1 should provide greater power than the t-test as it will account for the repeated observations of the endpoints over time. For Hypothesis 2, the investigators will look at one aspect of the feasibility of home-based practice as the ratio of those who achieve at least 150 minutes of weekly walking (composed of bouts that exceed 5 minutes) and 100 minutes of weekly upper extremity practice using the LEAP with the whole group as the denominator. The investigators anticipate that >75% will achieve this by the end of the intervention, based upon our preliminary studies using these devices in a chronic hemiparetic stroke population.

Secondary Analyses: Secondary outcomes listed in the Table will be evaluated using t-tests, Wilcoxon rank sum tests, or chi-square tests as appropriate. One planned secondary analysis will compare outcomes based on on whether or not participants can extend their wrist and at least 3 fingers at least 5 degrees at time of randomization, to assess for possible differences in drug responses between those with higher compared to lower levels of initial motor control. Another will compare outcomes in those who achieve the practice goals of Hypothesis 2 to those who do not in relation to drug assignment.

Safety Committee:

A Safety Committee will serve the research sites. It will include the study statistician, a physician and an allied health clinician with training in stroke rehabilitation. It will meet before the start of the trial, every 6 months, after the first 10 subjects have completed the 2-month drug intervention, and as needed (e.g., serious adverse reaction).

Confidentiality:

All data will be entered from both sites into the RedCap database that will be monitored at UCLA by the study statistician for completeness. All materials related to the trial for UCLA entries will be stored in a locked cabinet in a locked room by the coordinator.

ELIGIBILITY:
Inclusion Criteria:

* Transfer to inpatient rehabilitation within 4 weeks of stroke onset
* Single ischemic or subcortical hemorrhagic infarct;
* At the time of randomization, hemiparesis with 4/5 or less strength at the hip and ankle flexors and extensors
* Functional Independence Measure (FIM) score for ambulation ≥3 to walk at least 10 steps;
* Caregiver available for at least two hours a day for practice and transportation when needed;
* Adequate language skills to read and understand the Informed Consent and retain information during daily therapies.

Exclusion Criteria:

* Prior stroke with persisting motor impairment or disability;
* Limited resources or illness that will not enable a return to living outside of a facility;
* Any medical condition that had limited daily physical activity to walking no more than 2 blocks outdoors prior to the stroke (e.g., claudication, congestive heart failure or lower extremity pain);
* History of dementia or Mini Mental State Examination score <24;
* History of hepatitis or elevated hepatic transaminases or bilirubin;
* History of renal insufficiency or serum creatinine over 1.6;
* Cancer or other chronic illness that makes 3-year survival unlikely or will detract from the ability to carry out exercise and skills practice.

Ages: 30 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-10-01 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - California Rehabilitation Institute, Los Angeles, California
  - Yale University, New Haven, Connecticut
  - Burke Neurological Research Institute, White Plains, New York

RESULTS

PARTICIPANT FLOW:
Groups:
- Maraviroc + Augmented Rehabilitation: Maraviroc 300 mg daily for 60 days, plus receive rehabilitation therapy as prescribed by the doctors and via telerehabilitation.
- Placebo + Augmented Rehabilitation: Placebo 300 mg daily for 60 days, plus receive rehabilitation therapy as prescribed by the doctors and via telerehabilitation.
Period: Overall Study
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
Started | 2 | 0
8 Week Assessment | 0 | 0
6 Month Assessment | 0 | 0
Completed | 0 | 0
Not Completed | 2 | 0
Not completed — Withdrawal by Subject | 1 | 0
Not completed — COVID restrictions | 1 | 0

BASELINE CHARACTERISTICS:
Population: Only 2 participants were enrolled and began study activities before the study was halted prematurely due to recruitment difficulty.
Groups:
- Total: Total of all reporting groups
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 0 | 1
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 0 | 1
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 0 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 |  | 2

OUTCOME MEASURES:

1. Primary Outcome: Change in 10 Meter Walk Test
Description: Timed walking speed over 10 meters. The evaluable sample size of 30 in each group will have 80% power to detect a difference in means of -0.206 (m/s), the difference between an assumed usual care walking speed of 0.51 (SD=0.28) and an assumed intervention group mean walking speed of 0.716. This assumes a common standard deviation in the two groups and a two group t-test with a 0.05 two-sided significance level. The estimates for the mean and standard deviation for walking speed come from the LEAPS RCT (Duncan, N Engl J Med, 2011). The t-test used for the power calculation is a simplification of the mixed effects analysis plan for the primary endpoints.
Time Frame: Baseline, 6 months post
Population: Participants exited study prior to 6 month assessment
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Change in Action Research Arm Test
Description: Assessment of upper extremity function. Our sample size of 30 for each group is based on a statistical power of 80% with an alpha of 5% for detecting a meaningful difference of 6 points, i.e., a 10% change, which has been suggested by several completed trials. In a stroke trial, the standard deviation was 8 points measured at 2 weeks post stroke.
Time Frame: Baseline, 6 months post
Population: Participants exited study prior to 6 month assessment
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Fugl-Meyer Motor Score
Description: Assessment of arm and leg impairment after stroke
Time Frame: Baseline, within 5 days of last medication dose (8 weeks), at 6 months post stroke
Population: Participants exited study prior to 8 week assessment
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Stroke Impact Scale
Description: Self-report questionnaire on quality of life post-stroke
Time Frame: Baseline, within 5 days of last medication dose (8 weeks), at 6 months post stroke
Population: Participants exited study prior to 8 week assessment
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Change in 6 Minute Walking Distance
Description: Distance walked in a 6 minute time period
Time Frame: Baseline, within 5 days of last medication dose (8 weeks), at 6 months post stroke
Population: Participants exited study prior to 8 week assessment
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Change in Physical Activity Enjoyment Scale
Description: Self-report questionnaire related to exercise enjoyment
Time Frame: Baseline, within 5 days of last medication dose (8 weeks), at 6 months post stroke
Population: Participants exited study prior to 8 week assessment
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Change in Activity Self Efficacy
Description: Self-report questionnaire related to confidence in increasing activity and maintaining exercise routines
Time Frame: Baseline, within 5 days of last medication dose (8 weeks), at 6 months post stroke
Population: Participants exited study prior to 8 week assessment
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Change in International Physical Activity Questionnaire
Description: Self-report of activity levels
Time Frame: Baseline, within 5 days of last medication dose (8 weeks), at 6 months post stroke
Population: Participants exited study prior to 8 week assessment
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Change From Baseline in Walking Activity, Sensors
Description: Sedentary time
Time Frame: Collected daily for 8 weeks
Population: Participants exited study prior to assessment
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Upper Extremity Practice, Sensors
Description: Amount of time practicing
Time Frame: Collected daily for 8 weeks
Population: Participants exited study prior to complete assessment
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Upper Extremity Practice, Sensors
Description: Repetitions of task practice
Time Frame: Collected daily for 8 weeks
Population: Participants exited study prior to completion of assessment
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: No participants were enrolled in the Placebo arm prior to study termination
Arm/Group | Maraviroc + Augmented Rehabilitation | Placebo + Augmented Rehabilitation
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/0
Other Adverse Events (participants affected / at risk) | 0/2 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-08-01): https://cdn.clinicaltrials.gov/large-docs/26/NCT03172026/Prot_SAP_000.pdf